CLINICAL TRIAL: NCT07404995
Title: Analgesic Efficacy of Bilateral Erector Spinae Plane Block in Pediatric Tethered Cord Syndrome Surgery: A Prospective, Randomized Controlled Trial
Brief Title: Analgesic Efficacy of Bilateral Erector Spinae Plane Block in Pediatric Tethered Cord Syndrome Surgery
Acronym: ESPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, sermın emınoglu, ASSOCIATE PROFESSOR, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-KAEK-13
Record Dates: First submitted 2026-01-19; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Erector Spina Plan Block
Keywords: TETHERED CORD SENDROME; ESPB; TCI
MeSH Terms: interventions — Parapsychology; Dental Occlusion; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- UNDER ULTRASOUND GUİDANCE ESPB GROUP (Experimental): Under ultrasound guidance, bilateral erector spinae plane block will be performed on the ESPB group one level above the appropriate area for pediatric tethered cord surgery using the anesthetic drug bupivacaine.
  Interventions: Device: UNDER ULTRASOUND GUİDANCE ESPB BLOCK; Procedure: PROCEDURE/SURGERY: ERECTOR SPİNAE (ESP) BLOCK WİTH BUPİVACAİNE

INTERVENTIONS:
Device: UNDER ULTRASOUND GUİDANCE ESPB BLOCK — In the ESP Block group, with the patient in the prone position, the research anesthesia team will insert a block needle through the skin one level above the surgical level using a linear probe guided by USG. The needle will pass through the trapezius and erector spinae muscles, and upon reaching the transverse process (approximately 2-3 cm deep), a test dose of 0.5-1 mL of 0.9% NaCl will be applied between the erector spinae fascia and the vertebral transverse process to confirm needle placement. After confirmation of fascial opening, a local anesthetic volume of 2 mL per vertebral pressure will be calculated, not exceeding a maximum dose of 2 mg/kg of 0.5% bupivacaine. This total volume will be diluted by half with 0.9% NaCl solution to prepare a 0.25% bupivacaine concentration. The calculated local anesthetic solution will be applied to the erector spinae region for ESPB. The same procedures will be performed on the opposite side.
  Other Names: ESPB BLOCK
Procedure: PROCEDURE/SURGERY: ERECTOR SPİNAE (ESP) BLOCK WİTH BUPİVACAİNE — For the ESP Block group, under USG guidance with the patient in prone position, a linear probe will be placed in the parasagittal plane one level above the operative level, and after visualizing the transverse process with an in-plane approach, a 50 mm long block needle will be inserted through the skin. A test dose of 0.5-1 mL of 0.9% NaCl will be administered between the erector spinae fascia and the transverse process of the vertebra to confirm needle placement. After confirming that the fascia has opened, a local anesthetic volume of 2 mL per vertebral pressure will be calculated, not exceeding a maximum dose of 2 mg/kg of 0.5% bupivacaine. This total volume will be diluted halfway with 0.9% NaCl solution to prepare a 0.25% bupivacaine concentration. The calculated local anesthetic solution will be administered to the erector spinae area, and ESPB will be performed. The same procedures will be performed on the opposite side.
  Other Names: PLANE BLOCKS

SUMMARY:
Tethered Cord Syndrome is a developmental anomaly of neuroaxis characterized by stretching of the spinal cord and is diagnosed in the pediatric age group. Surgical release of the tight and tethered filum terminale is performed. Intraoperative neurophysiological monitoring (IONM) is used to preserve functional nerve tissue and prevent postoperative neurological deficits. Total intravenous anesthesia (TIVA-TCI) with propofol and remifentanil is used as the anesthesia method to ensure accurate measurements. Postoperative pain is acute pain caused by surgical trauma and signal transmission in afferent neurons. Pediatric postoperative pain is associated with adverse behaviors, prolonged hospital stay, and impaired functional recovery. Although good progress has been made in pain management, ineffective postoperative pain management in children remains a global problem. Regional anesthesia is increasingly used in pediatric patients to provide postoperative analgesia and support intraoperative anesthesia. Ultrasound-guided erector spinae plane block (ESPB) is a new approach. First introduced in 2016 by Forero et al., ESPB is a novel regional anesthesia technique that blocks the branches of spinal nerves by injecting a local anesthetic into the fascial plane between the erector spinae muscle and the transverse process. The aim of our study was to reduce intraoperative anesthetic drug consumption, postoperative pain levels in the first 24 hours, the need for analgesics, and unwanted side effects associated with analgesics by applying bilateral ESPB in pediatric patients operated on for Tethered Cord Syndrome. Our hypothesis in this study is that bilateral ESPB reduces intraoperative anesthetic drug consumption and the need for postoperative analgesia in pediatric patients operated on for Tethered Cord Syndrome.

DETAILED DESCRIPTION:
Ultrasound-guided erector spinae plane block (ESPB) that aims for the ventral and dorsal rami of the spinal nerves was recently introduced in spine surgery to treat postoperative pain. ESPB was reported to be effective in scoliosis surgery as it reduced the need for analgesic drugs. Due to its relative technical simplicity, the main advantages postulated for the ESPB are few complications and minimal risk for spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:Patients whose parents have given their consent to the study

* Patients aged 18 and under
* Patients with ASA (American Society of Anesthesiologists) physical status I, II, and III
* Pediatric patients who will undergo elective Tethered Cord Syndrome surgery

Exclusion Criteria:Patients whose parents did not consent to participate in the study

* Patients with ASA physical status IV and V
* Those using anticoagulant medications
* Allergy to local anesthetic drugs
* Patients with a history of gastrointestinal bleeding
* Those with infection in the area where the block is planned

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
INTRAOPERATİVE ANESTHETİC DRUG CONSUMPTİON BY APPLYİNG BİLATERAL ESPB İN PEDİATRİC PATİENTS. | İNTRAOPERATİVE
  TOTAL PROPOFOL (MİLLİGRAM) and TOTAL REMİFENTANYL (MİCROGRAM)

SECONDARY OUTCOMES:
POSTOPERATIVE PAIN SCORES | POSTOPERATIVE SERVICE 0. MINUTE 30.MINUTE 12.HOURS 5. MINUTE 1. HOURS 24. HOURS 10. MINUTE 2.HOURS 15. MINUTE 4. HOURS 20. MINUTE 6.HOURS
  POSTOPERATİVE PAİN SCORE (0: NONE, 100: VERY SEVERE)

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa yüksek ihtisas eğitim ve araştırma hastanesi BURSA, Bursa, Türkiye, Bursa, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study protocol and results can be shared.

REFERENCES:
- [Result] Ali Gado A, Alsadek WM, Ali H, Ismail AA. Erector Spinae Plane Block for Children Undergoing Cardiac Surgeries via Sternotomy: A Randomized Controlled Trial. Anesth Pain Med. 2022 Apr 19;12(2):e123723. doi: 10.5812/aapm-123723. eCollection 2022 Apr. PMID 35991776

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT07404995/Prot_SAP_000.pdf